CLINICAL TRIAL: NCT02910661
Title: TAKE-IT TOO: Teen Adherence in KidnEy Transplant, Improving Tracking To Optimize Outcomes (Stage 1)
Brief Title: Teen Adherence in KidnEy Transplant, Improving Tracking To Optimize Outcomes (Stage 1)
Acronym: TAKE-IT TOO
Status: Completed | Type: Observational
Sponsor: Beth Foster (Other)
Collaborators: University of Pittsburgh (Other); St. Louis Children's Hospital (Other); Seattle Children's Hospital (Other); St. Justine's Hospital (Other); The Hospital for Sick Children (Other); British Columbia Children's Hospital (Other); Temple University (Other); Université de Montréal (Other)
Responsible Party: Sponsor-Investigator, Beth Foster, Associate Professor of Pediatrics, McGill University Health Centre/Research Institute of the McGill University Health Centre
Organization: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Other Study IDs: 2017-1764
Record Dates: First submitted 2016-09-19; First posted 2016-09-22 (Estimated); Last update posted 2017-09-28 (Actual); Status verified 2017-09

CONDITIONS: Medication Adherence
Keywords: Kidney Transplantation
MeSH Terms: conditions — Medication Adherence | interventions — Focus Groups

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Patients: Focus groups (n=6-8/group) will be conducted at 4 sites selected to maximize racial diversity and to ensure availability of adequate numbers in each age group (Montreal (incl. the McGill University Health Centre (MUHC), Centre Hospitalier Universitaire-Ste. Justine & CHUM ), Pittsburgh, Seattle, and St. Louis). Separate focus groups will be conducted with patients clustered by patient age to maximize homogeneity in developmental stage. Purposive sampling will be employed to ensure that each focus group includes patients with combinations of characteristics that are likely to account for variation in perspectives, including the major racial and ethnic groups, both sexes, time since transplant, and level of adherence.
  Interventions: Other: Focus Group
- Parents: Focus groups (n=6-8/group) will be conducted at Pittsburgh & Seattle. Focus groups will be conducted with parents clustered by patient age (12-14 y. & 15- 17 y.)
  Interventions: Other: Focus Group
- Healthcare professionals: One focus group of healthcare professionals (HCP) representing the variety of multidisciplinary transplant team members at each center will be convened. We will aim for 4-8 HCP per group; however, the number will be dictated by the composition and size of the transplant team at each site. We expect variability in the organization of care across the 7 sites, which represent 2 countries and small to large program sizes; including all sites will capture this variability.
  Interventions: Other: Focus Group

INTERVENTIONS:
Other: Focus Group — Concurrently at each site, an experienced facilitator, having no direct affiliation with the clinical team, will use standardized stakeholder-specific, semi-structured scripts (designed with patient and parent collaborators) to conduct the patient, parent, and HCP focus groups. The TAKE-IT intervention will be described, and Simplemed e-pillbox shown, to all focus groups. Questions posed to the patient and parent focus groups will focus on 2 themes: the intervention and electronic monitoring. Example stakeholder-specific scripts to guide the discussions are appended. Each focus group will last ~90 min. and be audio-recorded. An observer will take field notes.

SUMMARY:
The overall goal of the Teen Adherence in KidnEy transplant Improving Tracking TO Optimize Outcomes (TAKE-IT TOO) study is to adapt the successful TAKE-IT intervention, aimed at improving medication adherence in adolescent kidney transplant, for use in 'real world' clinical care. The specific aims of Stage 1 of this study are: (1) To understand the needs and preferences of stakeholders (kidney transplant recipients, parents, and healthcare professionals (HCP)) in order to optimize the TAKE-IT intervention for 'real world' use.

DETAILED DESCRIPTION:
TAKE-IT TOO is a prospective, 3-stage, sequential study using user-centered design techniques throughout. This entry describes Stage 1of TAKE-IT TOO. In Stage 1 we will conduct focus groups (FG) to gather data about the needs and preferences of stakeholders to inform adaptation of the Teen Adherence in Kidney transplant Effectiveness of Intervention Trial (TAKE-IT) intervention and features of a novel e-pillbox and adherence-tracking website. The protocols for Stages 2 and 3 will be submitted separately.

ELIGIBILITY:
Inclusion Criteria:

* Patients: Prevalent kidney-only transplant recipients 12-24 y, ≥3 months post-transplant.
* Parents: Parents of prevalent kidney-only transplant recipients 12-17 y (followed in a participating transplant center). Parents will be eligible to participate even if their child does not participate.
* HCP: transplant healthcare professionals (including representatives from variety of disciplines typically involved in promoting medication adherence)

Exclusion Criteria:

* Patients: Individuals with significant neurocognitive disabilities limiting their ability to understand and participate in their own care. Multiorgan transplant recipients. Patient or parent unable to communicate in English or French (Montreal only)
* Parents: Parents of patients 18-24 years old will be excluded

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Representative groups of stakeholders (patients, parents and HCP) will be recruited from renal transplant centers representing two healthcare systems and a variety of program sizes: 3 in the United States (UPMC [which includes both adult and pediatric programs], Seattle Children's Hospital and St. Louis Children's Hospital), and 5 in Canada (MUHC, Ste-Justine Hospital (HSJ), Centre Hospitalier de l'Université de Montréal (CHUM), Vancouver's British Columbia Children's Hospital, and Toronto's Hospital for Sick Children).
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2017-03-28 (Actual); Primary Completion 2017-08-06 (Actual); Study Completion 2017-08-06 (Actual)

PRIMARY OUTCOMES:
Stakeholders' needs and preferences | 90 minutes
  needs and preferences of young kidney transplant recipients, their parents, and HCP regarding electronic monitoring and adherence interventions

CONTACTS AND LOCATIONS:
Overall Officials: Bethany J Foster, MD, MSCE, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre; Annette DeVito Dabbs, PhD, Principal Investigator — University of Pittsburgh
Locations (9):
- United States (4):
  - Children's Hospital St-Louis, St Louis, Missouri
  - Temple University, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Seattle Children's Hospital, Seattle, Washington
- Canada (5):
  - BC Children's Hospital, Vancouver, British Columbia
  - University of Toronto Hospital for Sick Children, Toronto, Ontario
  - Centre Hospitalier de l'Université de Montréal, Montreal, Quebec
  - CHU Ste-Justine, Montreal, Quebec
  - Montreal Children's Hospital of the MUHC, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Yes
Data generated will be available for use to other investigators in the research community. Data may be used for hypothesis testing, and to generate preliminary data in support of future research projects. A Data Sharing Committee, composed site investigators will review requests submitted for use of the data. If the request is approved, the appropriate data analysis will be performed and the results sent to the requesting investigator. Alternatively, depending on the request, it may be more appropriate to provide the requesting investigator with certain segments of the data. If this is the case, a file of the requested data (de-identified) will be provided to the investigator.